CLINICAL TRIAL: NCT00750698
Title: A Phase 2, Exploratory Study of Erlotinib and SNDX-275 in Patients With Non-small Cell Lung Carcinoma Who Are Progressing on Erlotinib
Brief Title: A Phase 2 Exploratory Study of Erlotinib and SNDX-275 in Participants With Non-small Cell Lung Carcinoma Who Are Progressing on Erlotinib
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to business reasons, enrollment on the study was halted and the study terminated. The decision to close enrollment was not due to any safety concern.
Sponsor: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNDX-275-0403
Record Dates: First submitted 2008-09-08; First posted 2008-09-10 (Estimated); Results first posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Non Small Cell Lung Cancer
Keywords: lung cancer; non small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — entinostat; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erlotinib-responsive (Experimental): Participants self-administered entinostat in combination with continued erlotinib self-administration.
  "Erlotinib-responsive" participants are those who progressed following either a complete or partial response to erlotinib or a period of stable disease lasting at least 3 months.
  Interventions: Drug: Entinostat; Drug: Erlotinib
- Erlotinib-nonresponsive (Experimental): Participants self-administered entinostat in combination with continued erlotinib self-administration.
  "Erlotinib-nonresponsive" participants are those who either progressed immediately during treatment with erlotinib (after at least 1 full cycle of erlotinib treatment) or had an objective response or period of stable disease lasting less than 3 months.
  Interventions: Drug: Entinostat; Drug: Erlotinib

INTERVENTIONS:
Drug: Entinostat — Entinostat (10 milligrams [mg] fixed dose orally [PO] every 2 weeks [Q2W]) on Days 1 and 15 of a 28-day cycle for up to 6 cycles
  Other Names: SNDX-275
Drug: Erlotinib — Erlotinib (150 mg PO QD) for up to six (6) 28-day cycles
  Other Names: Tarceva

SUMMARY:
To evaluate the tumor responses to SNDX-275 (entinostat) in combination with continued erlotinib in participants with non-small Cell Lung Carcinoma (NSCLC) who are progressing on erlotinib.

ELIGIBILITY:
Inclusion Criteria:

1. Cytologically or histologically confirmed NSCLC of stage IIIb (pleural effusion) or IV
2. Disease is progressing (either no response to treatment or subsequent relapse after an objective response) on erlotinib treatment, based on at least 2 scans (the last being within 4 weeks of study enrollment and can serve as the baseline scan for the participant's screening into the study)
3. Recovered from any toxicity associated with the most recent cancer treatment (no greater than grade 1 toxicity on Common Terminology Criteria for Adverse Events scale or to prior baseline condition)
4. At least 1 measurable lesion ≥ 20 millimeters (mm) by conventional computed tomography (CT) scan or ≥ 10 mm by spiral CT scan
5. Eastern Cooperative Oncology Group performance score of 0, 1, or 2 and life expectancy of at least 3 months
6. Paraffin-embedded tumor specimen available for correlative studies
7. Male or female over 18 years of age
8. Hemoglobin ≥ 9.0 grams/deciliter; platelets ≥ 75 x 10^9/liter (L); absolute neutrophil count ≥ 1.0 x 10^9/L without the use of hematopoietic growth factors
9. Coagulation tests within the normal range
10. Bilirubin and creatinine less than 2 times the upper limit of normal for the institution
11. Aspartate aminotransferase and alanine aminotransferase less than 3 times the upper limit of normal for the institution
12. Potassium, magnesium and phosphorus within the normal range for the institution (supplementation is permissible)
13. Willing to use accepted and effective methods of contraception during the study (both men and women as appropriate) and for 3 months after the last dose of entinostat
14. Participant or legally acceptable representative has granted written informed consent before any study-specific procedure (including special screening tests) is performed

Exclusion Criteria:

1. Prior stem cell transplant
2. Symptomatic central nervous system involvement
3. Prior treatment with an histone deacetylase inhibitor
4. Concurrent anticancer therapy, with the exception of radiotherapy for a non-target study lesion
5. Currently taking medication(s) on the prohibited medication list
6. Systemic chemotherapy or treatment with an investigational agent within 28 days before enrollment
7. Current use of valproic acid
8. Untreated or unstable brain metastases, or taken steroids for this condition within 4 weeks of study drug administration
9. Currently active second malignancy, or any malignancy within the last 5 years other than cured basal or squamous cell skin carcinoma, cervical carcinoma in situ, or superficial bladder cancer
10. Inability to swallow oral medications or a gastrointestinal malabsorption condition
11. Uncontrolled infection requiring intravenous antibiotics, antivirals, or antifungals, known human immunodeficiency virus infection, or active hepatitis B or C infection
12. Abnormal cardiac function as defined as clinically significant findings on electrocardiogram (multifocal premature ventricular complexes, ST-T wave changes consistent with myocardial infarction or acute ischemia, QTc greater than 500 milliseconds), tachycardia, or left ventricular ejection fraction less than 40% on multigated acquisition scan
13. Another serious or uncontrolled medical condition within 3 months of enrollment such as hypertension, diabetes mellitus, or suppressed immune system
14. Known hypersensitivity to benzamides
15. Morbid obesity
16. Women who are currently pregnant or breast-feeding
17. Participant is currently enrolled in (or completed within 28 days) another investigational drug study
18. Participant unavailable for on-study or follow-up assessments
19. Participant has any kind of medical, psychiatric, or behavioral disorder that places the participant at increased risk for study participation or compromises the ability of the participant to give written informed consent and/or to comply with study procedures and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-08; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Adjei, MD, Study Chair — Roswell Park Cancer Institute
Locations (5):
- United States (5):
  - Sharp Clinical Oncology Research, San Diego, California
  - University of Miami, Miami, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Roswell Park Cancer Institute, Buffalo, New York
  - Medical University of South Carolina, Charleston, South Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 8 of the 70 planned participants had been enrolled when the study was closed to further enrollment.
Groups:
- Erlotinib Responsive: Participants self-administered entinostat in combination with continued erlotinib self-administration.
  "Erlotinib-responsive" participants are those who progressed following either a complete or partial response to erlotinib or a period of stable disease lasting at least 3 months.
- Erlotinib Nonresponsive: Participants self-administered entinostat in combination with continued erlotinib self-administration.
  "Erlotinib-nonresponsive" participants are those who either progressed immediately during treatment with erlotinib (that is, after at least 1 full cycle of erlotinib treatment) or had an objective response or period of stable disease lasting less than 3 months.
Period: Overall Study
Arm/Group | Erlotinib Responsive | Erlotinib Nonresponsive
Started | 6 | 2
Received at Least 1 Dose of Study Drug | 6 | 2
Completed | 0 | 0
Not Completed | 6 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Progressive disease | 5 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Erlotinib Responsive | Erlotinib Nonresponsive | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Customized [Count of Participants; unit: Participants]
  18 to <45 | 1 | 0 | 1
  45 to <65 | 2 | 2 | 4
  65 to <75 | 3 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 5
  Male | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (Complete Response, Partial Response, or Stable Disease for at Least 3 Months
Time Frame: At least 3 months
Population: Due to halted enrollment, data was not collected for analysis of this outcome measure.
Arm/Group | Erlotinib Responsive | Erlotinib Nonresponsive
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Progression-free Survival Rate
Time Frame: Up to 4 months
Population: Due to halted enrollment, data was not collected for analysis of this outcome measure.
Arm/Group | Erlotinib Responsive | Erlotinib Nonresponsive
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) through approximately 8 months
Arm/Group | Erlotinib Responsive | Erlotinib Nonresponsive
Serious Adverse Events (participants affected / at risk) | 2/6 | 0/2
Other Adverse Events (participants affected / at risk) | 5/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib Responsive (N=6) | Erlotinib Nonresponsive (N=2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Hemolytic anemia (Blood and lymphatic system disorders) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib Responsive (N=6) | Erlotinib Nonresponsive (N=2)
Oedema peripheral (General disorders) | 2 | 2
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Decreased appetited (Metabolism and nutrition disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Fatigue (General disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1
Mucosal inflammation (General disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Aspartate aminotransferase increased (Infections and infestations) | 0 | 1
Asthenia (General disorders) | 1 | 0
Blepharitis (Eye disorders) | 1 | 0
Blood alkaline phosphatase increased (Infections and infestations) | 0 | 1
Breath odour (Gastrointestinal disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Haemorrhage urinary tract (Renal and urinary disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Phlebitis (Vascular disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Costovertebral angle tenderness (Renal and urinary disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Due to business reasons, enrollment on the study was halted and the study terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes